CLINICAL TRIAL: NCT05712031
Title: Clinical Evaluation of Combined Tooth-implant Supported Prosthesis: Controlled Prospective Clinical Study
Brief Title: Combined Tooth-implant Supported Prostheses
Acronym: CTISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ORHUN EKREN (Other)
Responsible Party: Sponsor-Investigator, ORHUN EKREN, Associate Professor, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Orhun ekren
Record Dates: First submitted 2023-01-14; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Dental Implant; Short Dental Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group2 (Experimental): Mandibular first or second premolar is combined with standard length(8-12mm) dental implants to support 3 unit Fixed Partial Dentures
  Interventions: Procedure: Insertion of 1 Nucleoss T4 dental implants in posterior mandible
- Group3 (Experimental): Mandibular first or second premolar is combined with short dental implants(5-6mm) to support 3 unit Fixed Partial Dentures
  Interventions: Procedure: Insertion of 1 Nucleoss T5 dental implants in posterior mandible
- Group1 (Active Comparator): Standard length (8-12mm) dental implants are inserted in posterior mandible replacing either first premolar and first molar or second premolar and second molar to support 3 unit fixed partial dentures.
  Interventions: Procedure: Insertion of 2 Nucleoss T4 dental implants posterior mandible

INTERVENTIONS:
Procedure: Insertion of 1 Nucleoss T4 dental implants in posterior mandible — Nucleoss T4 dental implants is combined with first or second premolar to support 3 unit fixed partial dentures
  Arms: Group2
Procedure: Insertion of 1 Nucleoss T5 dental implants in posterior mandible — Nucleoss T5 dental implants is combined with first or second premolar to support 3 unit fixed partial dentures
  Arms: Group3
Procedure: Insertion of 2 Nucleoss T4 dental implants posterior mandible — 2 freestanding Nucleoss T4 dental implants is used to support 3 unit fixed partial dentures
  Arms: Group1

SUMMARY:
The goal of this clinical study is to evaluate clinical performance of combined tooth-implant supported 3 unit fixed partial dentures in the posterior mandible and was to compare and evaluate them with the complications of 3 unit fixed partial dentures supported with free standing dental implants.The main question[s] it aims to answer are:

1.Is there any difference in terms of mechanical and biological complications as well as marginal bone level between free standing and combined tooth-implant supported 3 unit Fixed Partial Dentures in posterior mandible.

Participants will receive either 2 dental implants(Control group) or 1 standart length dental implants to be combine with abutment tooth or 1 short dental implant to be combine with abutment tooth for supporting 3 unit fixed partial dentures.

DETAILED DESCRIPTION:
Purpose: The aim of the study was to evaluate clinical performance of combined tooth-implant supported 3 unit fixed partial dentures in the posterior mandible and was to compare and evaluate them with the complications of 3 unit fixed partial dentures supported with free standing dental implants.

Material and methods: 78 partially edentulous patients in the posterior mandible (Kennedy 1 and Kennedy 2), age between 18-65 with no systemic disorders were recruited for the study (n=26). Group 1served as control group and received 2 dental implants for supporting 3 unit fixed partial dentures (FPD). In group 2 dental implants longer than 8 mm and in group 3 shorter than 8 mm were inserted to replace first or second molar combined with first or second premolar respectively to support cement retained 3 units FPD. Periapical radiographs were taken with parallel technique for evaluation of marginal bone resorption (CBL) and modified plaque index (MPI), bleeding index (BI) and sulcus depth of abutment teeth was recorded at the time of FPD insertion, 6 months after FPD insertion and annually. Abutment tooth intrusions, de-cementation of the restoration, porcelain chipping/delamination, framework fracture, abutment screw loosening, abutment and abutment screw fracture, implant fracture were also recorded as complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with no systemic disorders,
2. Partial edentulous in the posterior mandible unilaterally or bilaterally with maxillary arch fully dentate or have teeth and/or implant supported FPD,
3. At least 3 months of healing after tooth extraction on implant site,
4. Periodontally and endodontically healthy abutment tooth to be combined with implant,
5. Patients who have good oral hygiene habits,
6. Patients smoking less than 10 cigarettes/day,
7. More than 2mm of keratinized gingiva on implant site

Ages: 37 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | At baseline
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs
Marginal bone loss | 6 months
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs
Marginal bone loss | 1 year
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs
Marginal bone loss | 2 years
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs
Marginal bone loss | 3 years
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs
Marginal bone loss | 4 years
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs
Marginal bone loss | 5 years
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs
Marginal bone loss | 6 years
  Mesial and distal marginal bone loss around dental implants is measured by periodical radiographs

SECONDARY OUTCOMES:
Modified gingival index | At baseline
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Modified gingival index | 6 months
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Modified gingival index | 1 year
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Modified gingival index | 2 years
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Modified gingival index | 3 years
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Modified gingival index | 4 years
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Modified gingival index | 5 years
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Modified gingival index | 6 years
  The clinician evaluated bleeding around selected teeth using a periodontal probe and by giving scores between 0 and 3
Plaque index | At baseline
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3
Plaque index | 6 months
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3
Plaque index | 1 year
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3
Plaque index | 2 years
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3
Plaque index | 3 years
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3
Plaque index | 4 years
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3
Plaque index | 5 years
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3
Plaque index | 6 years
  the clinician evaluated plaque accumulation around selected teeth using a periodontal probe and by giving scores to buccal, lingual, mesial and distal surfaces between 0 and 3

CONTACTS AND LOCATIONS:
Overall Officials: ORHUN EKREN, PhD, Study Director — Cukurova University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meffert RM, Langer B, Fritz ME. Dental implants: a review. J Periodontol. 1992 Nov;63(11):859-70. doi: 10.1902/jop.1992.63.11.859. PMID 1453301
- [Background] Rameh S, Menhall A, Younes R. Key factors influencing short implant success. Oral Maxillofac Surg. 2020 Sep;24(3):263-275. doi: 10.1007/s10006-020-00841-y. Epub 2020 Apr 23. PMID 32323043
- [Background] Zarb GA, Lewis DW. Dental implants and decision making. J Dent Educ. 1992 Dec;56(12):863-72. PMID 1487588
- [Background] Al-Omiri MK, Al-Masri M, Alhijawi MM, Lynch E. Combined Implant and Tooth Support: An Up-to-Date Comprehensive Overview. Int J Dent. 2017;2017:6024565. doi: 10.1155/2017/6024565. Epub 2017 Mar 23. PMID 28424733
- [Background] de Paula GA, Silva GC, Vilaca EL, Cornacchia TM, de Magalhaes CS, Moreira AN. Biomechanical Behavior of Tooth-Implant Supported Prostheses With Different Implant Connections: A Nonlinear Finite Element Analysis. Implant Dent. 2018 Jun;27(3):294-302. doi: 10.1097/ID.0000000000000737. PMID 29521677
- [Background] Tsouknidas A, Giannopoulos D, Savvakis S, Michailidis N, Lympoudi E, Fytanidis D, Pissiotis A, Michalakis K. The Influence of Bone Quality on the Biomechanical Behavior of a Tooth-Implant Fixed Partial Denture: A Three-Dimensional Finite Element Analysis. Int J Oral Maxillofac Implants. 2016 Nov/Dec;31(6):e143-e154. doi: 10.11607/jomi.5254. PMID 27861651
- [Background] Hosny M, Duyck J, van Steenberghe D, Naert I. Within-subject comparison between connected and nonconnected tooth-to-implant fixed partial prostheses: up to 14-year follow-up study. Int J Prosthodont. 2000 Jul-Aug;13(4):340-6. PMID 11203652
- [Background] Naert IE, Duyck JA, Hosny MM, Van Steenberghe D. Freestanding and tooth-implant connected prostheses in the treatment of partially edentulous patients. Part I: An up to 15-years clinical evaluation. Clin Oral Implants Res. 2001 Jun;12(3):237-44. doi: 10.1034/j.1600-0501.2001.012003237.x. PMID 11359481
- [Background] Gunne J, Astrand P, Lindh T, Borg K, Olsson M. Tooth-implant and implant supported fixed partial dentures: a 10-year report. Int J Prosthodont. 1999 May-Jun;12(3):216-21. PMID 10635188
- [Background] Nickenig HJ, Schafer C, Spiekermann H. Survival and complication rates of combined tooth-implant-supported fixed partial dentures. Clin Oral Implants Res. 2006 Oct;17(5):506-11. doi: 10.1111/j.1600-0501.2006.01259.x. PMID 16958689
- [Background] Schwartz SR. Short Implants: An Answer to a Challenging Dilemma? Dent Clin North Am. 2020 Apr;64(2):279-290. doi: 10.1016/j.cden.2019.11.001. Epub 2020 Jan 2. PMID 32111268
- [Background] Benlidayi ME, Ucar Y, Tatli U, Ekren O, Evlice B, Kisa HI, Baksi U. Short Implants Versus Standard Implants: Midterm Outcomes of a Clinical Study. Implant Dent. 2018 Feb;27(1):95-100. doi: 10.1097/ID.0000000000000710. PMID 29303816
- [Background] Jung RE, Al-Nawas B, Araujo M, Avila-Ortiz G, Barter S, Brodala N, Chappuis V, Chen B, De Souza A, Almeida RF, Fickl S, Finelle G, Ganeles J, Gholami H, Hammerle C, Jensen S, Jokstad A, Katsuyama H, Kleinheinz J, Kunavisarut C, Mardas N, Monje A, Papaspyridakos P, Payer M, Schiegnitz E, Smeets R, Stefanini M, Ten Bruggenkate C, Vazouras K, Weber HP, Weingart D, Windisch P. Group 1 ITI Consensus Report: The influence of implant length and design and medications on clinical and patient-reported outcomes. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:69-77. doi: 10.1111/clr.13342. PMID 30328189